CLINICAL TRIAL: NCT00949819
Title: The UCLA ASCAP Project is an Observational, Longitudinal, and Open-ended Study Aimed at Establishing a Structured Program of Non-interventional Follow-up for Localized Prostate Cancer.
Brief Title: Active Surveillance for Cancer of the Prostate (ASCaP)
Acronym: ASCaP
Status: Recruiting | Type: Observational
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 11-002281
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Low risk; Gleason 6; Active surveillance
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, buffy coat, prostate tissue cores and urine.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- no treatment: Men with previously untreated, early stage prostate cancer.
  Interventions: Other: Active surveillance

INTERVENTIONS:
Other: Active surveillance — Serial, long term data collection and active surveillance

SUMMARY:
Active Surveillance (A.S.) of prostate cancer (CaP) is the systematic monitoring of men with low-risk, localized lesions, with curative treatment of those whose tumors show substantial progression. A.S. is different from Watchful Waiting (W.W.), which is the palliative treatment of men with progressive prostate cancer.

DETAILED DESCRIPTION:
This protocol is not designed as a formal clinical trial, but rather an observational protocol; no treatments and no randomization are included. Longitudinally, specimens and clinical data will be collected to provide information on the following:

* Imaging studies of the prostate
* Rates of curative intervention
* Measures of tumor recurrence/progression
* Disease specific survival
* Overall survival
* Clinical data to track Quality of Life

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the prostate.
2. Clinically localized prostate cancer: T1-2, NX or N0, MX or M0.
3. No previous treatment for prostate cancer (including hormonal therapy, radiation therapy, surgery, or chemotherapy).
4. Patient has elected Active Surveillance as preferred management plan for prostate cancer.
5. Patient consent has been obtained according to local Institutional Review Board .
6. Patient is accessible and compliant for follow-up.

Exclusion Criteria:

1. Unwillingness or inability to undergo serial prostate biopsy.
2. Overall life expectancy less than 2 years
3. Advanced prostate cancer

Ages: 30 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 462 (Estimated)
Dates: Start 2009-07-04 (Actual); Primary Completion 2027-07-05 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Discover and confirm clinical parameters that predict aggressive disease as defined by pre-specified histological, PSA, clinical criteria, or outcomes based on these variables. | Interim data analysis will be made every year

SECONDARY OUTCOMES:
Determine the clinical predictors of disease progression. Measure the recurrence-free, disease-specific, and overall survival of men on active surveillance for clinically localized prostate cancer. Determine factors that lead to active intervention | Interim data analysis will be done each year

CONTACTS AND LOCATIONS:
Overall Officials: Leonard S Marks, M.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No